CLINICAL TRIAL: NCT04541277
Title: A Phase II, Single Arm Study of Tislelizumab Combined With DNA Demethylation Agent +/- CAG Regimen in the Treatment of Patients With High-risk AML or AML Patients Older Than 60 Years of Age Who Are Unfit for Intensive Chemotherapy
Brief Title: Combined Inhibition of PD-1 and DNA Hypomethylating Agent +/- Chemotherapy in High-risk AML or Elderly Patients With AML Who Are Unfit for Intensive Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDCXG-RR&ELDER
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia, in Relapsed or Refractory; Acute Myeloid Leukemia, Elderly, Unfit; Acute Myeloid Leukemia With Positive Minimal Residual Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tislelizumab; Decitabine; Azacitidine; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab with DAN hypmethylation agent +/- chemotherapy (Experimental): Decitabine, 20 mg/m2/d, IV, on days 1-5; or Azacitidine, 75 mg/m2/d,SC, on days 1-7.
  Aclamycin hydrochloride, 20 mg/d, IV, on day 1, 3, and 5 (For relapse/resistance AML, on days 1-5.); or idarubicin hydrochloride,10 mg/d, IV, on day 1, 3, and 5.
  Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cytarabine,100 mg, IV, q12h/d. For patients with one of the following conditions, cytarabine,10 mg, SC, q12h/d: (1) There are obvious heart, lung, and kidney complications; (2) Bone marrow is hypoproliferative; (3) Age> 75 years old; (4) Age> 60 years old who are unfit for standard-dose chemotherapy.
  Recombinant human granulocyte colony stimulating factor injection, 5 μg/kg, SC, from day 0 to stop of chemotherapy after the WBC count exceeds 10.0×10^9/L; or Pegylated recombinant human granulocyte stimulating factor injection Liquid, 100 μg/kg, SC, on day 0.
  Tislelizumab,200 mg, IV, on the next day after chemotherapy was stopped.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab combined with DNA demethylation agent +/- CAG regimen
  Other Names: Decitabine; Azacitidine; Cytarabine; Idarubicin; Aclarithromycin; Recombinant Human Granulocyte Colony Stimulating Factor; Pegylated Recombinant Human Granulocyte Colony Stimulating Factor

SUMMARY:
This phase II trial studies how well tislelizumab combined with DNA hypomethylation agent +/- CAG regimen (cytarabine, idarubicin / Aclarithromycin, rhG-CSF/ PEG-rhG-CSF) work in treating patients with high-risk acute myeloid leukemia (AML) or AML patients older than 60 years of age who are unfit for standard-dose chemotherapy. The expressions of PD-1 and PD-L1 are increased in AML cells. However, blocking the immune checkpoint alone has limited efficacy as a single agent in highly proliferative leukemia cells. During the recovery period after cytotoxic chemotherapy, the activation of PD-1/PD-L1 pathway may be increased and DNA hypomethylation agents can also up-regulate PD-1, PD-L1 and PD-L2 in AML patients. The up-regulation and activation of above immune checkpoint molecules are related to chemotherapy resistance. Therefore, adding chemotherapy and epigenetic regulation agents to Immune checkpoint blockade therapy may work better through overcoming drug resistance in AML treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legally authorized representative must provide written informed consent.
2. Meet the diagnostic criteria for acute myeloid leukemia (AML) with positive minimal residual disease (MRD), excluding those patients who are MRD-positive or MRD recurrence after allogeneic hematopoietic stem cell transplantation (HSCT); or meet the diagnostic criteria for relapsed AML, excluding those experience relapsed within 2 months after HSCT from matched sibling donor or within 3 months after HSCT from alternative donor; or meet the diagnostic criteria for refractory AML, excluding those patients within 2 months after HSCT from matched sibling donor or those patients within 3 months after HSCT from alternative donor.
3. Bone marrow (BM) or peripheral blood (PB) leukemia cells were measured to express PD-L1 within 3 months of entering the study.
4. The toxic side effects of the last treatment should be restored.
5. Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
6. Creatinine =< 1.5 x upper limit of normal (ULN). Serum bilirubin =< 1.5 x ULN. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN.
7. Karnofsky Performance Scale Index => 70.
8. The expected survival period is at least 12 weeks.
9. Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (b-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use an effective contraception method during the study and for 23 weeks after the last dose of the study drug; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 31 weeks following the last dose of study drug.

Exclusion Criteria:

1. Patients with positive minimal residual disease (MRD) or MRD recurrence after HSCT; or patients who relapse or refractory within 2 months after HSCT from matched sibling donor or within 3 months after HSCT from alternative donor.
2. History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years.
3. Any major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy within 2 weeks prior to the first dose of the study drugs.
4. Patients with any other known concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes; cardiovascular disease including congestive heart failure New York Heart Association [NYHA] class III or IV, myocardial infarction within 6 months, and poorly controlled hypertension; chronic renal failure; or active uncontrolled infection) which, in the opinion of the investigator could compromise participation in the study.
5. Patients unwilling or unable to comply with the protocol.
6. Patients who are on steroids (> 10 mg/day or equivalent) or immune suppression medications.
7. Patients with autoimmune diseases (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]).
8. Patients with a history of inflammatory bowel disease such as Crohn's disease and ulcerative colitis.
9. Patients known to be positive for hepatitis B surface antigen expression or with active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months), or with known human immunodeficiency virus (HIV) infection.
10. Current therapy with other systemic anti-neoplastic or anti-neoplastic investigational agents.
11. Females who are pregnant or lactating.
12. Any grade of not controlled graft versus host disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 months post-treatment
  The percentage of subjects with complete remission (CR) and incomplete hematological recovery (CRi) within 2 medication cycles.

SECONDARY OUTCOMES:
The percentage of subjects with CR and CRi with negative minimal residual disease (MRD) within 2 cycles. | Up to 3 months post-treatment
Duration of Remission (DOR) | Up to 1 year post-treatment
  The time from first obtaining CR or CRi to relapse or death from AML.
Progression-free survival time (PFS) | Up to 1 year post-treatment
  the time from the day of treatment to relapse, progression or death (whichever occurs first is preferred).
Overall survival (OS) | Up to 1 year post-treatment
  The time from the day of treatment to death.
28-day response rate | Up to 35 days post-treatment
  The percentage of subjects with CR and CRi (calculated based on the best response) at the 28th day after treatment.
Incidence of adverse events | Up to 35 days post-treatment
  The incidence of adverse events will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
PD-L1 expression in acute myeloid leukemia bone marrow cells | Up to 1 year post-treatment
  The expression levels of PD-L1 in acute myeloid leukemia bone marrow cells will be assessed at the 28th day after each medication cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Dai-hong Liu, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou HS, Su YF, Wang J, Hu YL, Wang A, Xu L, Wang YZ, Zheng X, Li YQ, Min KL, Gao CJ, Liu DH, Gao XN. Updates from a single-center phase 2 study of PD-1 inhibitor combined with hypomethylating agent plus CAG regimen in patients with relapsed/refractory acute myeloid leukemia. Front Immunol. 2025 Apr 17;16:1533467. doi: 10.3389/fimmu.2025.1533467. eCollection 2025. PMID 40313949
- [Derived] Gao XN, Su YF, Li MY, Jing Y, Wang J, Xu L, Zhang LL, Wang A, Wang YZ, Zheng X, Li YF, Liu DH. Single-center phase 2 study of PD-1 inhibitor combined with DNA hypomethylation agent + CAG regimen in patients with relapsed/refractory acute myeloid leukemia. Cancer Immunol Immunother. 2023 Aug;72(8):2769-2782. doi: 10.1007/s00262-023-03454-y. Epub 2023 May 11. PMID 37166484